CLINICAL TRIAL: NCT03697239
Title: Phase IB/II Trial of High Dose Ascorbic Acid (AA) + Nanoparticle Paclitaxel Protein Bound + Cisplatin + Gemcitabine (AA NABPLAGEM) in Patients Who Have No Prior Therapy for Their Metastatic Pancreatic Cancer
Brief Title: High Dose Ascorbic Acid (AA) + Nanoparticle Paclitaxel Protein Bound + Cisplatin + Gemcitabine (AA NABPLAGEM) in Patients Who Have Metastatic Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: FDA indicated the same study could not be conducted under multiple INDs
Sponsor: Hitendra Patel (Other)
Collaborators: Cancer Research UK (Other); Stand Up To Cancer (Other); Lustgarten Foundation (Other); Destroy Pancreatic Cancer (Other); Translational Genomics Research Institute (Other); HonorHealth Research Institute (Other)
Responsible Party: Sponsor-Investigator, Hitendra Patel, Associate Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 181045
Record Dates: First submitted 2018-09-21; First posted 2018-10-05 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Metastatic Pancreatic Cancer; Pancreatic Cancer; Pancreas Cancer; Pancreatic Adenocarcinoma Resectable; Pancreatic Ductal Adenocarcinoma; Pancreatic Metastasis
Keywords: metastatic pancreatic cancer; cancer; pancreatic; Vitamin C; Ascorbic Acid; Nanoparticle Paclitaxel Protein Bound; cisplatin; gemcitabine; pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Ascorbic Acid; Taxes; Cisplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Ascorbic Acid Paclitaxel Protein Bound Cisplatin Gemcitabine
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AA NABPLAGEM (Experimental): ascorbic acid paclitaxel protein-bound cisplatin gemcitabine
  Interventions: Drug: Ascorbic Acid; Drug: Paclitaxel protein-bound; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Ascorbic Acid — 25, 37.5, 56.25 or 75 grams/m2
  Other Names: Vitamin C
Drug: Paclitaxel protein-bound — 125mg/m2 over 30 minute IV infusions on days 1 and 8 repeated every 21 days
Drug: Cisplatin — 25mg/m2 in 500*mL of NS over 60minute IV infusion on days 1 and 8 repeated every 21 days
Drug: Gemcitabine — 1000mg/m2 in 500*mL over 30 minute IV infusion on days 1 and 8 repeated every 21 days

SUMMARY:
The purpose of this study is to see if a combination of paclitaxel protein bound (also known as nab-paclitaxel), gemcitabine, and cisplatin when given with high dose Ascorbic Acid will be safe and effective in individuals with untreated metastatic pancreatic cancer.

Vitamin C is a nutrient found in food and dietary supplements. It protects cells and also plays a key role in making collagen (which provides strength and structure to skin, bones, tissues and tendons). High-dose vitamin C may be given by intravenous (IV) infusion (through a vein into the bloodstream) or orally (taken by mouth). When taken by intravenous infusion, vitamin C can reach much higher levels in the blood than when the same amount is taken by mouth. Some human studies of high-dose IV vitamin C in patients with cancer have shown improved quality of life, as well as improvements in physical, mental, and emotional functions, symptoms of fatigue, nausea and vomiting, pain, and appetite loss. Intravenous high-dose ascorbic acid has caused very few side effects in clinical trials.

DETAILED DESCRIPTION:
Pancreatic cancer continues to be a very lethal disease. It was estimated that in 2016, 53,070 Americans would be diagnosed with pancreatic ductal adenocarcinoma (PDA), and 41,780 would die from the disease. This makes pancreatic cancer the third leading cause of death from cancer in the US.

PDA is the twelfth most common cancer in the world with 338,000 new cases diagnosed in 2012. It is estimated that worldwide there will be > 300,000 deaths from pancreatic cancer. Furthermore unfortunately PDA is projected to be the second leading cause of death from cancer in the US by 2030.

Detection of pancreatic cancer has notoriously been very late in the disease and therefore the 5-year survival rate is only 8%, which is actually a slight improvement over the last few years. Right now the only potential cure for pancreatic cancer is surgical resection (if the disease is caught early). However only about 20% of PDA patients are eligible for potentially curable resection and unfortunately most (> 80%) have recurrence of their cancer within 2 years of resection, and those recurrences are almost universally fatal.

Recently it has been shown that there are regimens that actually improve survival for patients with advanced stage IV PDA. Conroy and colleagues have developed the Folfirinox regimen, which in a large randomized trial improved survival over gemcitabine as a single agent. Von Hoff and colleagues developed the nanoparticle albumin (nab) associated paclitaxel plus gemcitabine regimen which improved survival over single agent gemcitabine. Even more recently Jameson and colleagues have presented a combined regimen of nab-paclitaxel + gemcitabine + cisplatin in a small 24 patient phase Ib/II trial which showed a response rate of 71% with 2 patients having complete response, a 1-year survival of 65% and a median survival of 16+ months.

While there have been multiple investigators and investigations into the use of ascorbic acid for patients with cancer (see ClinTrials.gov), its use has generally not been found to be of help for patients particularly when given orally - e.g. 10 grams daily.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma (with measurable disease according to RECIST 1.1 criteria).
* Adequate organ function

Exclusion Criteria:

* Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatments in the adjuvant setting with gemcitabine and/or 5-FU or gemcitabine administered as a radiation sensitizer are allowed, provided at least 6 months have elapsed since completion of the last dose
* Palliative surgery and/or radiation treatment less than 4 weeks prior to initiation of study treatment.
* Exposure to any investigational agent within 4 weeks prior to initiation of study treatment.
* Patients who need constant use of finger stick blood glucose monitoring for tight control of their diabetes
* Any person with a G6PD deficiency
* History of renal oxalate stones
* Patient is taking acetaminophen at any dose, or any medication that contains acetaminophen within 72 hours of first dose of ascorbic acid.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Is pregnant or breastfeeding
* Current, serious, clinically significant cardiac arrhythmias or receiving a digitalis derivative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 18 weeks
  To determine the maximum tolerated dose (MTD) of high dose ascorbic acid (AA) with triple therapy of nanoparticle paclitaxel protein bound + cisplatin + gemcitabine (NABPLAGEM) in patients with advanced stage IV metastatic pancreatic cancer
Disease Control Rate | 18 weeks
  CR+ PR+SD

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Grade 2-5 Adverse Events assessed using NCI CTCAE v5.0 toxicity criteria | 18 weeks
Percent of patients who normalize their CA19-9 | 18 weeks
  Lab testing will be completed to evaluate normalization of CA19-19
Progression free survival (PFS) | approximately 12 weeks from last study treatment
  Telephone follow up will be conducted every 12 weeks from the last dose of treatment to determine status of disease progression
Overall survival (OS) | approximately 12 weeks from last study treatment
  Telephone follow up will be conducted every 12 weeks from the last dose of treatment to determine survival status
Changes in patient's self-reported quality of life | 18 weeks
  Changes in patient's self-reported quality of life will be determined by administering the MD Anderson Symptom Inventory (MDASI-GI)
Changes in patient's self-reported pain levels | 18 weeks
  Changes in patient's self-reported quality of life will be determined by administering the MD Anderson Symptom Inventory (MDASI-GI)

CONTACTS AND LOCATIONS:
Overall Officials: Hitendra Patel, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States